CLINICAL TRIAL: NCT05768659
Title: Implicit Reactions to Threats in Individuals With Obesity: Primary Evidence From Fear Conditioning Paradigm
Brief Title: Fear Conditioning Paradigm in Obesity
Acronym: GenAllertOB
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21X101
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: fear conditioning; fear processing; anxiety
MeSH Terms: conditions — Obesity; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Participants affected by obesity (the level of body mass index (BMI) higher or equal to 30).
  Interventions: Behavioral: Fear Conditioning
- Controls: Not-hospitalized participants with a healthy weight
  Interventions: Behavioral: Fear Conditioning

INTERVENTIONS:
Behavioral: Fear Conditioning — It is a 2-day paradigm. Participants will undergo an auditory fear conditioning task in 3 phases: (1) pre-conditioning habituation, (2) unconditioned stimulus (US) calibration, where USs will be delivered to set the individual stimulation intensity threshold, and (3) fear conditioning, in which participants will be exposed to the conditioned stimulus (CS) associated with the US with an 80% pairing rate. 24 hours later, the (1) implicit recognition of the CS and novel stimuli (NSs), and the (2) explicit recognition, through an alternative forced-choice task will be assessed. Also, (3) the perceptual discrimination (among the CS and NSs) will be tested.
  Event-related skin conductance responses (SCRs) will be collected as an implicit index of defensive fear responses, while the accuracy in detecting and discriminating the CS from NSs as the explicit index. Psychological questionnaires about anxiety symptoms will be also administered.

SUMMARY:
Fear processing in obesity and specifically the ability to i) learn and remember threatening stimuli, and ii) implicitly (i.e., unconsciously) and explicitly (consciously) discriminate them from neutral ones, will be investigated in affected individuals through the fear-conditioning paradigm.

ELIGIBILITY:
Inclusion criteria:

* Right-handed
* diagnosis of obesity (the level of body mass index - BMI - higher or equal to 30).

Exclusion criteria:

• concurrent neurological, neurodevelopmental (e.g., autism), motor, somatosensory and/or psychiatric disorders.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with obesity will be recruited at the beginning of a rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy). Controls will be recruited out of the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
SCRs) | Baseline
  The event-related skin conductance responses (SCRs) in the case of the CS will be measured. This will represent the implicit index.

SECONDARY OUTCOMES:
Recognition % | baseline
  Level of accuracy (in %) in recognizing and discriminating the CS from NS will be computed. This will represent the explicit index.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano - Ospedale San Giuseppe, Piancavallo, VCO, Italy